CLINICAL TRIAL: NCT06663462
Title: EzPAP Therapy Versus Non-invasive Ventilation for Hypercapnic Chronic Obstructive Pulmonary Disease Exacerbataion: a Randomized Clinical Trial
Brief Title: EzPAP Therapy Versus Non-invasive Ventilation Therapy
Status: Completed | Type: Observational
Sponsor: Kırklareli University (Other)
Responsible Party: Principal Investigator, Oya Guven, MD, Assistant Professor, Kırklareli University
Other Study IDs: Training and Research Hospital
Record Dates: First submitted 2024-10-19; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Non Invasive Ventilation
Keywords: Chronic Obstructive Pulmonary dissease; Non-invasive ventilation; EzPAP

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EzPAP group: EzPAP users
- Non-invasive group: BPAP users

SUMMARY:
This study compared EzPAP and noninvasive treatments of hypercapnic COPD attacks.

DETAILED DESCRIPTION:
In this study, the effectiveness of NIV and EzPAP treatments was compared in patients admitted to the emergency department due to hypercapnic COPD exacerbation. Blood gas was taken at the 4th and 24th hours of treatment to evaluate the effectiveness.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Chronic obstructive pulmonary disease Dyspnea

Exclusion Criteria:

Cardiac failure Dead

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD disease
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Blood gas | 24 hours
  Carbon dioxide height, low bicarbonate and presence acidosis measure in the blood gas

CONTACTS AND LOCATIONS:
Overall Officials: Gökhan Karakurt, MD, Study Director — Kırklareli Training and Research Hospital
Locations (1):
- Oya Guven, MD, Kırklareli, Center, Turkey (Türkiye)